CLINICAL TRIAL: NCT06839118
Title: Safety and Efficacy of Botulinum Toxin A in Patients With Posttraumatic Headache: a Double-blind, Randomized, Placebo-controlled, Parallel-group Trial and Investigation of Neuroinflammatory Biomarkers as Predictors of Efficacy
Brief Title: Safety and Efficacy of Botulinum Toxin A in Patients With Posttraumatic Headache
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Henrik Schytz, Associate Professor, Danish Headache Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-515901-24-00
Record Dates: First submitted 2025-02-03; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Posttraumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BTX-A (Experimental): BTX-A used in this study will be Botox® and delivered in vials. A concentration of 50U/mL BTX-A is prepared using saline in four syringes: one with 1 mL, one with 0.8 mL, one with 0.7 mL, one with 0.6 mL. This equals a total administration dose of 155U.
  Interventions: Drug: Botox 200 UNT Injection
- Isotonic saline (Placebo Comparator): Placebo syringes are prepared exclusively with similar amounts of fluid as in the BTX-A arm.
  Interventions: Drug: Botox 200 UNT Injection

INTERVENTIONS:
Drug: Botox 200 UNT Injection — A concentration of 50U/mL BTX-A is prepared using saline in four syringes: one with 1 mL, one with 0.8 mL, one with 0.7 mL, one with 0.6 mL. This equals a total administration dose of 155U. A total of 155U BTX-A will be injected at day 1 (first day in week 1) by subcutaneous injections according to the PREEMPT protocol.
  Other Names: Botulinumtoxin-A

SUMMARY:
The study is an investigator-initiated randomized, placebo-controlled, double-blind, parallelgroup trial. Eighty subjects with PTH will be included and randomized 1:1 for treatment with BTX-A or placebo (isotonic saline). The study comprises a 4-week baseline phase before injection of either active drug or placebo followed by a 12-week evaluation period. Treatment will be double-blind, and subjects will only receive one treatment cycle. Endpoints will be assessed in the evaluation period (weeks 5 to 8) compared to baseline (weeks -4 to -1).

DETAILED DESCRIPTION:
Post-traumatic headache (PTH) accounts for 4% of all symptomatic headache disorders and is one of the most common consequences of mild traumatic brain injury, also known as concussion. There is significant overlap between PTH and primary headache disorders, making treatment strategies highly dependent on the specific headache pattern.

Initial treatment typically involves common analgesics, with triptans as an alternative option. For patients experiencing persistent PTH or inadequate response to acute treatment, preventive medication is recommended based on the characteristics of their headache. While PTH is classified as a secondary headache disorder, its symptoms often resemble migraine, suggesting a potential overlap in underlying molecular mechanisms.

One molecule that has drawn attention in this context is calcitonin gene-related peptide (CGRP), which plays a key role in migraine pathogenesis. Studies have shown that intravenous infusion of CGRP can trigger migraine attacks, while CGRP antagonism has been effective for both acute and preventive migraine treatment. Supporting its role in PTH, research has indicated that blocking CGRP may have therapeutic benefits for patients with persistent PTH. Additionally, animal studies have suggested that concussed rodents exhibit hypersensitivity to CGRP, further implicating its involvement in post-traumatic headache.

The relationship between botulinum toxin type A (BTX-A) and CGRP has also been explored in experimental models using capsaicin. Capsaicin activates sensory nerve fibers, causing pain through the release of pain mediators such as CGRP and substance P. Interestingly, BTX-A has been shown to reduce pain, inflammation, and hyperalgesia by blocking CGRP release, which may contribute to its clinical effectiveness.

Botulinum Toxin A (BTX-A) BTX-A is a neurotoxin produced by Clostridium botulinum that inhibits the release of acetylcholine at the neuromuscular junction, leading to muscle relaxation. When administered subcutaneously to the face and scalp, BTX-A has been approved as a preventive treatment for chronic migraine, as well as several other conditions.

In the treatment of trigeminal neuralgia, BTX-A is used off-label, with injections of 50-150 units in affected areas supplied by branches of the trigeminal nerve. The treatment is generally well-tolerated, with minimal side effects, such as mild muscle weakness at the injection site. Importantly for PTH, BTX-A does not cause cognitive side effects. However, scientific evidence supporting its effectiveness in PTH remains weak, and well-powered randomized controlled trials are needed.

Research suggests that BTX-A can reduce inflammation in the periosteum and inhibit the release of signaling molecules such as CGRP. It also prevents the insertion of pain-related ion channels in the synaptic membrane, which are involved in pain processing. Additionally, CGRP and vasoactive intestinal peptide (VIP) have been identified as potential biomarkers predicting the effectiveness of BTX-A in other pain conditions. BTX-A has also been shown to decrease inflammatory biomarkers, including interleukin-1 at the trigeminal ganglion and tumor necrosis factor alpha in experimental pain models. These findings suggest that BTX-A may act as a modulator of neuronal signaling and neuroinflammation, providing a potential mechanism for its effect in treating PTH.

Clinical Efficacy and Safety of BTX-A The effectiveness of BTX-A was evaluated in a study involving 40 PTH patients who were randomly assigned to receive either BTX-A or a saline placebo. The study assessed changes in headache frequency, severity, and the number of headache days per week. Patients treated with BTX-A experienced a significant reduction in weekly headaches, with a decrease of 2.24 headaches per week (43.3%). In contrast, those receiving placebo experienced an increase of 1.28 headaches per week (35.1%). The difference between the two groups was statistically significant, supporting the potential benefit of BTX-A for PTH treatment.

Rationale for Study Endpoints During the evaluation period, the primary measure of efficacy in this study is the change in the number of moderate-to-severe headache days compared to baseline. A moderate-to-severe headache day is defined as a day with headache pain of moderate or severe intensity lasting at least 30 minutes without medication or a headache that responds to acute treatment. A clinically meaningful treatment response is considered to be a reduction of at least 30% in moderate-to-severe headache days.

Rationale for Injection Site and Dosage Patients will receive 155 units of BTX-A through 31 injections of 5 units each, following the PREEMPT protocol. The placebo will consist of isotonic saline administered through 31 injections of 0.1 ml each.

Investigating Neuroinflammatory Biomarkers There is limited research on neuroinflammatory biomarkers and their role in PTH. This study could provide valuable insights into the underlying mechanisms of PTH and determine whether biomarkers can predict treatment response. Since the trigeminal nerve innervates the cornea, measuring CGRP levels in tear fluid may be a more sensitive method for detecting concentration changes compared to blood plasma, given the tear fluid's proximity to trigeminal nerve endings.

Clinical Hypothesis BTX-A reduces the number of moderate-to-severe headache days in PTH patients with minimal side effects, making it an effective and safe treatment.

In PTH patients, changes in neuroinflammatory biomarker concentrations are significantly greater in those who respond to BTX-A compared to non-responders or those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of persistent PTH according to criteria 5.2.2 Persistent headache attributed to mild traumatic injury to the head according to The International Classification of Headache Disorders 3rd edition.
2. Age between 18 and 80 years.
3. Subjects must have headache at least 15 days per month during the last 4 weeks to enter the baseline phase.
4. During baseline phase subjects must experience moderate-to-severe headache at least 8 days and headache at least 15 days to enter the treatment phase (to be randomized).
5. Fluency in Danish

Exclusion Criteria:

1. More than 2 TBI's.
2. Severe cardiovascular and cerebrovascular disease such as ischemic heart disease, myocardial infarction or previous stroke or transient ischemic attack, major CVD interventions during the last three months.
3. Expected poor compliance, i.e., considered unlikely to be able to complete all protocol required study visits or procedures, and/or to comply with all required study procedures to the best of the subject's and investigator's knowledge.
4. Ongoing and unstable severe psychiatric disease.
5. Anamnestic or clinical symptoms of any kind that are deemed relevant for study participation by the physician who examines the patient.
6. A history of migraine or tension-type headache more than 5 days per month before the TBI.
7. Medication-overuse headache according to the according to The International Classification of Headache Disorders 3rd edition.
8. A history of moderate-to-severe TBI, whiplash injury, or craniotomy.
9. Change of preventive PTH treatment or treatment dose within two months prior to the baseline visit (see Section 6.4 for a full list of these medications).
10. Previous treatment with injections of BTX-A in the head or face.
11. Female subjects either pregnant, breastfeeding or with planned conception within the study period.
12. Female subject of childbearing potential who is unwilling to use an acceptable method of effective contraception during the study. Acceptable methods of effective birth control include not having intercourse (true abstinence, when this is in line with the preferred and usual lifestyle of the subject), hormonal birth control methods (pills, shots/injections, implants, or patches), intrauterine devices, surgical contraceptive methods (vasectomy with medical assessment of the surgical success of this procedure or bilateral tubal ligation). Female subjects not of childbearing potential are defined as any female who: is post-menopausal by history, defined as:

    1. Age ≥ 55 years with cessation of menses for 12 or more months, OR
    2. Age < 55 years but no spontaneous menses for at least 2 years, OR
    3. Age < 55 years and spontaneous menses within the past 1 year, but currently amenorrheic (e.g., spontaneous, or secondary to hysterectomy), AND with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved OR underwent bilateral oophorectomy OR underwent hysterectomy OR underwent bilateral salpingectomy.
13. Known allergy to any component of BTX-A.
14. Infection at the proposed injection site.
15. Known severe neuromuscular disorders or any degree of disorder affecting the neuromuscular transmission.
16. Known comprised respiratory function.
17. Member of investigational site staff or relative of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Primary aim | 3 months
  To investigate if botulinum toxin type A (BTX-A) is safe and more effective than placebo to lower the number of moderate-to-severe headache days in the evaluation period (weeks 5 to 8) compared to baseline (weeks -4 to -1). Headache days will defined as mild, moderate or severe in intensity based on the International Headache Society guideline for conduction studies on preventive medication in post-traumatic headache

SECONDARY OUTCOMES:
First secondary aim | 2 months
  To investigate the degree of change in inflammatory biomarkers concentration in plasma and tears in responders versus non-responders in the BTX-A and placebo groups at week 0 and week 8.
Second secondary aim | 3 months
  To investigate the proportion of subjects reaching a ≥50% or a ≥75% reduction in the number of days with moderate-to-severe headache during the evaluation period (weeks 5 to 8) compared with baseline (weeks -4 to -1), respectively.
Third secondary aim | 3 months
  To evaluate the change from baseline period (weeks -4 to -1) to evaluation period (weeks 5 to 8) in Headache Impact Test (HIT-6) at week 8 in the BTX-A group versus the placebo group.
Fourth secondary aim | 3 months
  To evaluate the change from baseline period (weeks -4 to -1) to evaluation period (weeks 5 to 8) in Headache Impact Test (HIT-6) at week 8 in the BTX-A group versus the placebo group.
Fifth secondary aim | 3 months
  To evaluate the effectiveness of blinding. Participants will be asked to guess which study drug was administered to make sure that blinding was not broken because of visible discrete facial paralysis.
Sixth secondary aim | 3 months
  To evaluate tolerability and safety by A. Evaluating the proportion of dropouts caused by increased intake of posttraumatic headache (PTH) medication or use of prohibited rescue medication in the BTX-A group compared to the placebo group. B: Evaluating the proportion of subjects with side effects registered in the evaluation period (weeks 5 to 8) in the BTX-A group compared to the placebo group.
Seventh secondary aim | 3 months
  To evaluate the change from baseline period (weeks -4 to -1) to evaluation period (weeks 5 to 8) in Rivermead Post-Concussion Symptoms Questionnaire at week 8 in the BTX-A group versus the placebo group.
Eight secondary aim | 3 months
  To evaluate the change from baseline period (weeks -4 to -1) to evaluation period (weeks 5 to 8) in Hospital Anxiety and Depression Scale (HADS) at week 8 in the BTX-A group versus the placebo group.
Ninth secondary aim | 3 months
  To evaluate the change from baseline period (weeks -4 to -1) to evaluation period (weeks 5 to 8) in The Insomnia Severity Index (ISI) at week 8 in the BTX-A group versus the placebo group.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No